CLINICAL TRIAL: NCT07403214
Title: Disease-modifying Therapies (DMT) Treatment Outcomes in Patients With Spinal Muscular Atrophy (SMA) - A Real-world Study Using the Komodo Claims Data
Brief Title: A Real-world Study of Disease-modifying Therapy Treatment Outcomes in Patients With Spinal Muscular Atrophy
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COAV101A1US09
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Muscular Atrophy, Spinal
Keywords: Spinal muscular atrophy; Multiple disease modifying therapies; Real-world evidence; Treatment patterns
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (8):
- DMT Cohort A: Patients with SMA who were treated with at least 1 DMT and had continuous health insurance coverage in KRD+ closed claims at the time of first DMT initiation.
- DMT Cohort B: Patients with SMA who were treated with at least 1 DMT and received the first DMT at age 2 or younger.
- DMT Cohort B1: A sub-group of DMT Cohort B who started the first DMT between 2016 and 2021.
- DMT Cohort B2: A sub-group of DMT Cohort B who started the first DMT between 2022 and 2024.
- DMT Cohort C: Patients with SMA types 1-3 who were treated with multiple DMTs.
- DMT Cohort D: A subset of DMT Cohort C who received the first DMT at age two or younger.
- DMT Cohort D1: A sub-group of DMT Cohort D who started the first DMT between 2016 and 2021.
- DMT Cohort D2: A sub-group of DMT Cohort D who started the first DMT between 2022 and 2024.

SUMMARY:
The aim of this study was to evaluate treatment patterns, SMA-related complications and services, and all-cause medical encounters of patients with SMA receiving multiple DMTs in the real world. The DMTs included onasemnogene abeparvovec-xioi (OA), nusinersen, and risdiplam. This study was conducted using data from the Komodo Health Research Database (KRD+) between 01 January 2016 and 31 October 2024.

ELIGIBILITY:
Inclusion criteria

* Patients with ≥1 SMA diagnosis at any time (International Classification of Disease, Tenth Revision, Clinical Modification [ICD-10-CM] codes: G12.0, G12.1, G12.9).
* Patients with ≥1 record of OA, nusinersen, or risdiplam based on relevant Healthcare Common Procedure Coding System (HCPCS) codes and National Drug Code (NDC).
* Patients who received at least 2 of the 3 DMTs, with the first DMT initiated on or after 26 May 2019, when at least 2 DMTs were available. The initiation of the first DMT was defined as the index date and the first DMT was defined as the index DMT.
* Patients with SMA types 1, 2, or 3.
* Patients with ≥1 quarter of clinical activities within 1 year prior to the index quarter (for patients with SMA type 2 and 3 only).
* Patients with ≥1 quarter of clinical activities any time after the index quarter, unless death occurred.

Exclusion criteria

* Patients with SMA type 4.
* Patients with claims of multiple DMTs in their birth year.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SMA patients with data in the KRD+ between 01 January 2016 and 31 October 2024 who received OA, nusinersen, or risdiplam.
Sampling Method: Non-Probability Sample
Enrollment: 4805 (Actual)
Dates: Start 2025-06-04 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Patients by SMA-related Complication, Procedure, and Durable Medical Equipment (DME) Before Receiving the First DMT (Period I) | Up to approximately 1 year
  DME is medical equipment that assists patients with their medical condition, can be used at home, and lasts a long time.
Number of Patients by SMA-related Complication, Procedure, and DME After Receiving the First DMT and Before the Second DMT (Period II) | Up to an average of approximately 2 years
  DME is medical equipment that assists patients with their medical condition, can be used at home, and lasts a long time.
Number of Patients by SMA-related Complication, Procedure, and DME After Receiving the Second DMT and Before the Third DMT (Period III) | Up to an average of approximately 2 years
  DME is medical equipment that assists patients with their medical condition, can be used at home, and lasts a long time.
Number of Patients by All-cause Medical Encounters During Period I | Up to approximately 1 year
  Medical encounters included outpatient visits, inpatient admissions, emergency room visits, and specialist visits.
Number of Patients by All-cause Medical Encounters During Period II | Up to an average of approximately 2 years
  Medical encounters included outpatient visits, inpatient admissions, emergency room visits, and specialist visits.
Number of Patients by All-cause Medical Encounters During Period III | Up to an average of approximately 2 years
  Medical encounters included outpatient visits, inpatient admissions, emergency room visits, and specialist visits.
Number of Medical Encounters per Patient per Year (PPPY) During Period I | Up to approximately 1 year
  Medical encounters included outpatient visits, inpatient admissions, emergency room visits, and specialist visits.
Number of Medical Encounters PPPY During Period II | Up to an average of approximately 2 years
  Medical encounters included outpatient visits, inpatient admissions, emergency room visits, and specialist visits.
Number of Medical Encounters PPPY During Period III | Up to an average of approximately 2 years
  Medical encounters included outpatient visits, inpatient admissions, emergency room visits, and specialist visits.
Inpatient Visit Length of Stay PPPY During Period I | Up to approximately 1 year
Inpatient Visit Length of Stay PPPY During Period II | Up to an average of approximately 2 years
Inpatient Visit Length of Stay PPPY During Period III | Up to an average of approximately 2 years

SECONDARY OUTCOMES:
Number of Patients who Received Multiple DMTs by Order in Which DMTs were Received | Up to approximately 5 years and 5 months
Time Between the First and Second DMT Initiation Among Patients Treated With Multiple DMTs | Up to an average of approximately 2 years
Time Between the Second and Third DMT Initiation Among Patients Treated With Multiple DMTs | Up to an average of approximately 2 years
Time on the First DMT During Period II Among Patients Treated With Multiple DMTs | Up to an average of approximately 2 years
Time on the First DMT During Period III Among Patients Treated With Multiple DMTs | Up to an average of approximately 2 years
Time on the Second DMT During Period III Among Patients Treated With Multiple DMTs | Up to an average of approximately 2 years
Number of Patients who Started a Second DMT | Up to approximately 5 years and 5 months
Duration of Continuous Enrollment for Patients Treated With at Least 1 DMT | Up to approximately 5 years and 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No